CLINICAL TRIAL: NCT07191795
Title: Uses of Phantom Sensations Induced by Global and Local Modifications of the Prosthetic Socket as Somatosensory Feedback During Walking in Lower Limb Amputees
Acronym: PhantomWalk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Collaborators: Clinique Chantecler (Unknown); Centre Orthopédique Maguelone (Unknown); Centre Helio Marin (Unknown); Institut universitaire de réadaptation Valmante Sud (Unknown); Institut des Sciences du Mouvement (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-A01647-36; ANR-23-CE17-0067-02 (Other: ANR)
Record Dates: First submitted 2025-08-21; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lower Limb Amputation
Keywords: Phantom Limb Sensation; Referred Sensation; Somatosensory Feedback; Lower Limb Prosthesis; Prosthetic Gait
MeSH Terms: interventions — Gait Analysis; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TT (Experimental): People with transtibial amputation
  Interventions: Other: Gait analysis; Other: Mapping of referred sensations.; Other: Phantom limb interview
- TF (Experimental): People with transfemoral amputation
  Interventions: Other: Gait analysis; Other: Mapping of referred sensations.; Other: Exploration of the areas of the brain activated during referred sensations; Other: Evaluation of the effects of socket modifications on phantom sensations and walking; Other: Phantom limb interview
- Control (Experimental): Asymptomatic people
  Interventions: Other: Gait analysis; Other: Exploration of the areas of the brain activated during referred sensations

INTERVENTIONS:
Other: Gait analysis — Participants with unilateral amputations and a control group will undergo a comprehensive walking analysis. In a lab setting (on a treadmill or floor), their gait will be recorded using inertial sensors, EMG, force plates, and motion capture, while an EEG cap and a NASA-TLX questionnaire will assess cognitive load. Capable participants will also perform a walking test on a real-world outdoor course with varied terrain. The data will be analyzed to compare walking patterns between groups (amputees vs. controls, and amputees with vs. without phantom limbs). Finally, participants will describe any interactions they perceived between their phantom sensations and walking during the tests.
Other: Mapping of referred sensations. — Participants reporting referred sensations in gait analysis phase will undergo further testing. The study will investigate whether prosthesis pressure or a specific socket interaction causes these sensations. A 3x3 cm grid will be drawn on the residual limb to systematically map referred sensations using various stimuli (brush, pressure tip, electrical stimulation). Participants will rate the intensity and describe the location of any resulting phantom sensations. This mapping will be repeated after 6 months to assess the stability of these sensations over time, with the ultimate goal of potentially using them to provide sensory feedback for prosthesis users. The session will last approximately 2 hours.
  Arms: TF; TT
Other: Exploration of the areas of the brain activated during referred sensations — Unilateral transfemoral amputees with detailed referred sensation maps will have their brain activity recorded using a 64-electrode EEG cap. Non-invasive stimuli will be applied to four specific sites: an area on the residual limb that elicits a referred sensation, the corresponding location on the intact foot, a neutral area on the residual limb, and its corresponding location on the intact thigh. This process, involving 400 total stimulations, will be repeated after 6 months to track cortical changes. Non-amputee participants will also be tested as a control group to check for symmetry in brain responses to thigh stimulation. Each session lasts about 2 hours.
  Arms: Control; TF
Other: Evaluation of the effects of socket modifications on phantom sensations and walking — This phase will evaluate how socket modifications affect phantom sensations and walking in 10 transfemoral amputees. First, the best material to comfortably induce referred sensations will be determined in a small sub-study. Then, each participant will be tested under four conditions: their usual socket and a socket with different rigidity, both with and without a specific local pressure point added inside. The location of this pressure point is based on the user's sensation map. Participants' walking will be analyzed in both lab and real-world environments for each condition, and they will provide feedback on their sensations and which setup they find most helpful. The evaluation involves 4 sessions over 2-3 months
  Arms: TF
Other: Phantom limb interview — A semi-structured interview will be conducted to ask participants to describe their phantom limb sensations (type, location, intensity) under three conditions: without their prosthesis, while standing with it, and while walking with it. This aims to identify factors influencing these sensations. Additionally, a brief physical examination of the residual limb will be performed to see if touch in specific areas triggers any referred sensations.
  Arms: TF; TT

SUMMARY:
Following lower-limb amputation, the loss of somatosensory information from the missing limb renders walking less automatic, more cognitively demanding, and often asymmetric, which can lead to secondary pathologies.

Hypothesis: This study is based on the hypothesis that phantom limb sensations (PLS), when coherent with the prosthetic device's movements and the phases of the gait cycle, can compensate for the loss of somatosensory feedback and thereby improve locomotion for individuals with amputation. It is further hypothesized that it is possible to artificially induce these coherent and useful sensations, notably through "referred sensations" elicited by stimulation of the residual limb (e.g., via the prosthetic socket).

Objectives: The project aims to:

* Determine whether the natural presence of phantom limb sensations during walking impacts gait parameters.
* Confirm in a larger patient population that modifications to the prosthetic socket can induce or enhance phantom sensations that are perceived as useful for walking.
* Investigate whether these perceptual changes (induced or enhanced) are associated with objective, measurable improvements in gait quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants with amputations:

  * Major lower limb amputation
  * Understand and be able to express oneself in the French language (for semi-structured interviews)
  * Affiliated with a social security scheme
* Asymptomatic volunteer participants:

  * No major surgery on the lower limbs for at least 3 years
  * No minor injury to the trunk, lower or upper limbs that could influence walking for at least 1 year
  * Understand and be able to express oneself in the French language
  * Affiliated with a social security scheme

Exclusion Criteria:

* History of psychiatric disorders
* Pregnant or breastfeeding woman
* Minor
* Adult subject to a legal protection measure
* Person under guardianship or conservatorship
* Person under a judicial protection order
* Pain affecting walking (trunk, residual limb, phantom limb, contralateral limb)
* Medical treatment incompatible with walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of phantom limb sensations | The first day of the study
  A composite assessment of phantom limb sensations will be conducted via a semi-structured interview. Data collected will include:
  * Type of sensation (e.g., tingling, pain, movement).
  * Location (toes, heel, calf).
  * Intensity (Mild, Strong, Very Strong).
Walking speed under laboratory conditions | The first day of the study for the control group and the second day of the study for participants with amputation
  The participant's average walking speed, measured in meters per second (m/s). The measurement will be collected using inertial measurement units (IMUs) and/or a Vicon motion capture system while the participant walks on hard ground or on a treadmill at their self-selected speed.
Step length symmetry index. | The first day of the study for the control group and the second day of the study for participants with amputation
  Gait symmetry will be calculated based on the stride length of the affected (or corresponding) limb and the healthy limb. The symmetry index is a unitless ratio (or percentage) that quantifies the difference between the two limbs. A value of 1 (or 100%) indicates perfect symmetry. Measured using inertial measurement units or the Vicon system.
Changes in the surface area of sensory maps referred to the residual limb | 2nd or 3rd day of the study depending on whether the participant with an amputation was included in phase 2 or not and during the 6-month follow-up visit.
  The total surface area capable of triggering phantom sensations will be measured. For each type of stimulation (brush, pressure, point, electrical), the number of 3x3 cm areas causing a sensation will be counted. The total surface area (in cm²) will be calculated by multiplying this number by 9. A map will be generated for each stimulation modality.
Change in the average intensity of reported phantom sensations. | 2nd or 3rd day of the study depending on whether the participant with an amputation was included in phase 2 or not and during the 6-month follow-up visit.
  When each reactive area is stimulated, the participant will rate the intensity of the phantom sensation perceived on a 6-point Numerical Rating Scale (NRS), ranging from 0 (no sensation) to 5 (maximum intensity imaginable). The average intensity of the reactive areas will be calculated for each type of stimulation.
Localization of the cortical source of somatosensory evoked potentials (SEPs) during stimulation of referred sensation areas | The second day of the study for participants with amputation
  The recorded EEG activity will be used to model and locate the source of the maximum cortical response. The primary outcome measure will be the coordinates (e.g., in the MNI or Talairach atlas) of the center of activation in the somatosensory cortex. The objective is to compare the source localization obtained during ecological gait after each demanding walking situation.
Participant's subjective preference for one of the four socket conditions tested. | Day 7 of the study
  At the end of the four test sessions, participants will be asked to rank the four conditions (rigidity A/B, with/without focal pressure) from most to least conducive to walking. The primary outcome will be the condition ranked first by the largest number of participants.
Change in the spatiotemporal parameters of walking in ecological situations | Days 4 to 7 to the study
  Several key walking parameters (speed in m/s, cadence in steps/min, step symmetry index) will be measured using inertial sensors during the outdoor walk. The analysis will compare the average values of these parameters between the four socket conditions.

SECONDARY OUTCOMES:
Walking pace under laboratory conditions | The first day of the study for the control group and the second day of the study for participants with amputation
  The number of steps per minute (steps/min) when walking at a comfortable speed. Measured using inertial measurement units or the Vicon system.
Analysis of muscle co-activation in the lower limbs and trunk during walking. | The first day of the study for the control group and the second day of the study for participants with amputation
  The electrical activity of key muscle groups (e.g., quadriceps, hamstrings, glutes, paravertebral muscles) will be recorded using surface electromyography (EMG). The analysis will focus on the timing and amplitude of muscle activation to assess motor coordination.
Maximum vertical reaction force during walking. | The first day of the study for the control group and the second day of the study for participants with amputation
  The maximum force exerted on the ground with each step, measured in Newtons (N) or as a percentage of body weight (%BW). The measurement will be taken using force platforms (AMTI), pressure insoles (Loadsol), or an instrumented mat (Zeno).
Assessment of mental workload during walking using the NASA-TLX questionnaire | The first day of the study for the control group and the second day of the study for participants with amputation
  The cognitive load perceived by the participant will be assessed using the NASA Task Load Index (NASA-TLX) self-report questionnaire. The total score, ranging from 0 to 100, will be calculated. A higher score indicates a greater perceived cognitive load.
Analysis of brain activity related to cognitive load during walking | The second day of the study for participants with amputation
  Electroencephalographic (EEG) activity will be recorded via a headset. Cognitive load will be quantified by analyzing the power ratio in specific frequency bands at the frontal electrodes.
Gait speed in ecological situation | The first day of the study for the control group and the second day of the study for participants with amputation
  The average walking speed (in m/s) measured using inertial measurement units and pressure soles (Loadsol) during a predefined outdoor route including various difficulties (stairs, slopes, etc.).
Qualitative description of the interaction between phantom sensations and walking | The second day of the study for participants with amputation
  Participants' verbal descriptions of the nature of the interaction (facilitating, hindering, neutral), the evolution and characteristics of phantom sensations during walking will be collected via a structured interview at the end of the session. The data will be analyzed thematically.
Change in phantom limb sensation intensity at 6 months for recent amputees | The first day of the study and during the 6-month follow-up visit.
  For the subgroup of participants with an amputation of less than 6 months at inclusion, the intensity of phantom sensations will be re-assessed using the 3-point ordinal scale.
Effect of focal stimulation on phantom sensations | Day 3 of the study
  For the subgroup of participants reporting interaction between sensations and focal stimulation after various stimulations using a rubber tip (pressure), a brush, and a needle. The change in sensation intensity (rated on a scale of 0 to 5). The result will be categorized as "increase," "decrease," or "no change."
Change in perceived cognitive load (NASA-TLX score) during walking in an ecological setting | Day 4 to 7 of the study
  Perceived mental workload will be assessed using the NASA-TLX questionnaire immediately after each walking session. The total score will be compared between the four socket conditions.
Evaluation of socket comfort | Day 4 to 7 of the study
  The overall comfort perceived for each condition will be assessed at the end of each session using a Numerical Rating Scale (NRS) ranging from 0 (very uncomfortable) to 10 (very comfortable). The average score will be compared between the four conditions.
Qualitative description of the sensations reported for each socket condition | Day 4 to 7 of the study
  For each condition, a structured description of the sensations reported (type, location, intensity, perceived usefulness for walking) will be collected through an interview. The data will be analyzed thematically to compare the sensory experience.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie A Touillet, Principal Investigator — Institut Régional de Médecine Physique et de Réadaptation
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France